CLINICAL TRIAL: NCT03219424
Title: Predicting the Probability of Return to Work After Injury in Hong Kong: Prospective Multicentre Cohort Study
Brief Title: Predicting the Probability of Return To Work After Injury
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: CREC2016.667-T
Record Dates: First submitted 2017-07-07; First posted 2017-07-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Trauma
Keywords: Return to work status; Functional outcome; Quality of life
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate return to work (RTW) status after moderate and major trauma in Hong Kong at one year after injury. To derive reliable prediction models for return to work.

DETAILED DESCRIPTION:
Background:

Trauma is a leading cause not only of death worldwide but also of disability, and in Hong Kong it ranks sixth as a cause of death for all age groups. The implementation of trauma systems has improved the survival of injured patients in many settings including Hong Kong. However, the aim of trauma care for the injured person is not only to prolong life but also to restore patients to the best possible health status, and where applicable, to return to work. Survivors of trauma often experience late sequelae that have a major impact on almost all aspects of everyday life, and improvements in functional outcome and health status may continue for at least five years post-injury.

Objectives:

1. to evaluate return to work (RTW) status after moderate and major trauma in Hong Kong at one year after injury;
2. to derive reliable prediction models for RTW.

Study design:

This is a multi-centre, prospective long-term follow up cohort study of the 1163 trauma patients admitted to the Prince of Wales Hospital (PWH), Queen Elizabeth Hospital (QEH) and Tuen Mun Hospital (TMH) in Hong Kong in 2017-2018. Patients will be recruited within four weeks of ED attendance as soon as the patient is clinically stable and conscious. The follow-up period for return to work status of the 1163 trauma patients will extend from baseline to one year after trauma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Eligible for the trauma registry
* Working or seeking employment before injury

Exclusion Criteria:

* Isolated hip or pathological fractures
* Injury severity score (ISS) of 1
* Patients who are unwilling to enter the study
* Patients who have left Hong Kong

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients aged 18 years or above who enter into the trauma registry of the hospitals involved in the study between 1 September 2017 and 31 August 2018 inclusive will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1115 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Return to work status at 12 months after injury | 12 months after injury
  The proportion of trauma patients who return to work at 12 months after injury

SECONDARY OUTCOMES:
Change of Glasgow Outcome Scale-Extended (GOSE) over time | On admission, 30 days after injury, 3 months after injury, 6 months after injury, 9 month after injury and 12 months after injury
  Change of GOSE over time

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung KKC, Leung LY, Yeung JHH, Wong TK, Yiu TY, Leung YK, Chan LPS, Wong JKS, Leung MPS, Goggins WB, Chan DYC, Lui CT, Ng WK, Ho HF, Cheng CH, Cheung NK, Graham CA. Return to work after injury in Hong Kong: prospective multi-center cohort study. Eur J Trauma Emerg Surg. 2022 Aug;48(4):3287-3298. doi: 10.1007/s00068-022-01899-x. Epub 2022 Feb 17. PMID 35175362